CLINICAL TRIAL: NCT01728376
Title: A Comparative Evaluation of the Safety and Efficacy of Daptomycin Versus Standard of Care in Pediatric Subjects One - Seventeen Years of Age With Bacteremia Caused by Staphylococcus Aureus.
Brief Title: Safety & Efficacy of Daptomycin Versus Standard of Care (SOC) in 1 - 17 Year Olds With Staphylococcus Aureus Bacteremia (MK-3009-005)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cubist Pharmaceuticals LLC, a subsidiary of Merck & Co., Inc. (Rahway, New Jersey USA) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3009-005; DAP-PEDBAC-11-02 (Other: Cubist Pharmaceuticals LLC Protocol Number)
Record Dates: First submitted 2012-11-05; First posted 2012-11-19 (Estimated); Results first posted 2016-12-07 (Estimated); Last update posted 2018-08-28 (Actual); Status verified 2018-07

CONDITIONS: Bacteremia
MeSH Terms: conditions — Bacteremia | interventions — Daptomycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Daptomycin - 12 to 17 year olds (Experimental): Participants ages 12-17 years old were administered daptomycin 7 mg/kg infused once daily, intravenously (IV), over 30 minutes; therapy duration (uncomplicated bacteremia) = 5-28 days, therapy duration (complicated bacteremia) = 7-42 days. After conclusion of IV therapy, can continue on oral therapy (not daptomycin, but at discretion of investigator).
  Interventions: Drug: Daptomycin
- Comparator - 12 to 17 year olds (Active Comparator): Participants ages 12-17 years old received IV vancomycin or semi-synthetic penicillin or first-generation cephalosporins or clindamycin, given as per local guidelines or site-specific prescribing information; therapy duration (uncomplicated bacteremia) = 5-28 days, therapy duration (complicated bacteremia) = 7-42 days. IV comparator and subsequent oral therapy were at the discretion of the investigator.
  Interventions: Drug: Comparator
- Daptomycin - 7 to 11 year olds (Experimental): Participants ages 7 to 11 years old were administered daptomycin 9 mg/kg, infused once daily, IV over 30 minutes; therapy duration (uncomplicated bacteremia) = 5-28 days, therapy duration (complicated bacteremia) = 7-28 days. After conclusion of IV therapy, can continue on oral therapy (not daptomycin, but at discretion of investigator).
  Interventions: Drug: Daptomycin
- Daptomycin - 1 to 6 year olds (Experimental): Participants ages 1 to 6 years old were administered daptomycin 12 mg/kg, infused once daily, IV over 60 minutes; therapy duration (uncomplicated bacteremia) = 5-28 days, therapy duration (complicated bacteremia) = 7-28 days. After conclusion of IV therapy, can continue on oral therapy (not daptomycin, but at discretion of investigator).
  Interventions: Drug: Daptomycin
- Comparator - 7 to 11 year olds (Active Comparator): Participants ages 7-11 years old received IV vancomycin, or semi-synthetic penicillin, or first-generation cephalosporins, clindamycin; given as per local guidelines or site-specific prescribing information; therapy duration (uncomplicated bacteremia) = 5-28 days, therapy duration (complicated bacteremia) = 7-28 days. IV comparator and subsequent oral therapy were at the discretion of the investigator.
  Interventions: Drug: Comparator
- Comparator - 1 to 6 year olds (Active Comparator): Participants ages 1-6 years old received IV vancomycin, or semi-synthetic penicillin, or first-generation cephalosporins, clindamycin; given as per local guidelines or site-specific prescribing information; therapy duration (uncomplicated bacteremia) = 5-28 days, therapy duration (complicated bacteremia) = 7-28 days. IV comparator and subsequent oral therapy were at the discretion of the investigator.
  Interventions: Drug: Comparator

INTERVENTIONS:
Drug: Daptomycin — Intravenous daptomycin given at 7 mg/kg (ages 12-17 years); 9 mg/kg (ages 7-11 years); 12 mg/kg (ages 1-6 years) infused once daily, intravenously, over 30 or 60 minutes. Participants may be switched to oral therapy following completion of IV study drug administration provided they showed clear clinical improvement and the pathogen was susceptible to an oral agent.
  Other Names: Cubicin
  Arms: Daptomycin - 1 to 6 year olds; Daptomycin - 12 to 17 year olds; Daptomycin - 7 to 11 year olds
Drug: Comparator — Vancomycin, Semi-synthetic penicillin, First-generation cephalosporins, Clindamycin: administered per standard of care. Participants may be switched to oral therapy following completion of IV study drug administration provided they showed clear clinical improvement and the pathogen was susceptible to an oral agent.
  Arms: Comparator - 1 to 6 year olds; Comparator - 12 to 17 year olds; Comparator - 7 to 11 year olds

SUMMARY:
The intent of this study is to describe the safety and efficacy of daptomycin versus standard of care (SOC) in pediatric participants aged 1-17 years with bacteremia caused by Staphylococcus aureus (S. aureus).

DETAILED DESCRIPTION:
S. aureus causes a series of invasive diseases in adults and children, including bacteremia. Infections due to S. aureus in children, particularly those due to methicillin resistant S. aureus (MRSA), are a growing world-wide public health concern.

Daptomycin, a cyclic lipopeptide antibacterial agent, shows rapid in vitro bactericidal activity with concentration-dependent killing for Gram-positive organisms, including S. aureus. Surveillance studies have demonstrated a daptomycin MIC90 of 0.5µg/ml for both methicillin-susceptible S. aureus (MSSA) and MRSA with >99% of MRSA isolates being categorized as susceptible by the Food and Drug Administration (FDA), European Committee of antimicrobial susceptibility testing (EUCAST) and Clinical and Laboratory Standards Institute (CLSI) breakpoints (5). Clinical trials in adults demonstrated that daptomycin was safe and efficacious in complicated skin and skin structure infections (cSSSI) and bloodstream infections caused by S. aureus, including right-sided infective endocarditis (RIE). However, information on the safety and efficacy of daptomycin for use in children is lacking.

The intent of this study in children is to confirm the safety of daptomycin at mean steady state systemic exposures (AUC) similar to those reported for adults treated at 6 mg/kg for bacteremia.

ELIGIBILITY:
Inclusion Criteria:

To be included in this study, participants must:

* Sign a parental consent form; if appropriate, sign an assent form
* Be between 1 and 17 years of age
* Have proven or probable bacteremia caused by S. aureus based on the traditional culture result, rapid diagnostic test or Gram stain
* If female of childbearing potential, must not be pregnant or nursing and take appropriate measures to not get pregnant during the study
* If male, must take appropriate measures to not get partner pregnant
* Able to comply with the protocol requirements

Exclusion Criteria:

Participants will not be allowed into the study if they:

* Have received a certain amount of antibacterial therapy specific for current bacteremia unless it is demonstrated that the organism is resistant to the given antibacterial;
* Anticipate to require other antibiotics that may be potentially effective against S. aureus;
* Have shock or hypotension unresponsive to standard therapy;
* Have received an investigational product or have participated in an experimental procedure within 30 days;
* Have an intolerance or hypersensitivity to daptomycin;
* Have renal insufficiency;
* Have prior history or current evidence of muscle damage (rhabdomyolysis; significant CPK elevation);
* Have history of clinically significant muscular disease, nervous system or seizure disorder, including unexplained muscular weakness, history of peripheral neuropathy, Guillain-Barré or spinal cord injury;
* Have S. aureus pneumonia, empyema, meningitis, or endocarditis

Ages: 1 Year to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 82 (Actual)
Dates: Start 2012-11-29 (Actual); Primary Completion 2016-01-20 (Actual); Study Completion 2016-01-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Derived] Arrieta AC, Bradley JS, Popejoy MW, Bensaci M, Grandhi A, Bokesch P, Glasser C, Du L, Patino H, Kartsonis NA. Randomized Multicenter Study Comparing Safety and Efficacy of Daptomycin Versus Standard-of-care in Pediatric Patients With Staphylococcal Bacteremia. Pediatr Infect Dis J. 2018 Sep;37(9):893-900. doi: 10.1097/INF.0000000000001926. PMID 29406465

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants aged 1-17 with bacteremia caused by Staphylococcus aureus (S. aureus) were enrolled in this study.
Groups:
- Daptomycin - 1 to 6 Year Olds: Participants ages 1 to 6 years old were administered daptomycin 12 mg/kg, infused once daily, intravenously (IV) over 60 minutes; therapy duration (uncomplicated bacteremia) = 5-28 days, therapy duration (complicated bacteremia) = 7-28 days. After conclusion of IV therapy, can continue on oral therapy (not daptomycin, but at discretion of investigator).
- Comparator- 1 to 6 Year Olds: Participants ages 1-6 years old received IV vancomycin, or semi-synthetic penicillin, or first-generation cephalosporins, clindamycin; given as per local guidelines or site-specific prescribing information; therapy duration (uncomplicated bacteremia) = 5-28 days, therapy duration (complicated bacteremia) = 7-28 days. IV comparator and subsequent oral therapy were at the discretion of the investigator.
- Daptomycin - 7 to 11 Year Olds: Participants ages 7-11 years old were administered daptomycin 9 mg/kg infused once daily, intravenously, over 30 minutes; therapy duration (uncomplicated bacteremia) = 5-28 days, therapy duration (complicated bacteremia) = 7-28 days. After conclusion of IV therapy, can continue on oral therapy (not daptomycin, but at discretion of investigator).
- Comparator - 7 to 11 Year Olds: Participants ages 7-11 years old received IV vancomycin or semi-synthetic penicillin or first-generation cephalosporins or clindamycin, given as per local guidelines or site-specific prescribing information; therapy duration (uncomplicated bacteremia) = 5-28 days, therapy duration (complicated bacteremia) = 7-28 days. IV comparator and subsequent oral therapy were at the discretion of the investigator.
- Daptomycin - 12 to 17 Year Olds: Participants ages 12-17 years old were administered daptomycin 7 mg/kg infused once daily, intravenously, over 30 minutes; therapy duration (uncomplicated bacteremia) = 5-28 days, therapy duration (complicated bacteremia) = 7-42 days. After conclusion of IV therapy, can continue on oral therapy (not daptomycin, but at discretion of investigator).
Period: Overall Study
Arm/Group | Daptomycin - 1 to 6 Year Olds | Comparator- 1 to 6 Year Olds | Daptomycin - 7 to 11 Year Olds | Comparator - 7 to 11 Year Olds | Daptomycin - 12 to 17 Year Olds | Comparator - 12 to 17 Year Olds
Started | 22 | 11 | 19 | 9 | 14 | 7
Treated | 22 | 10 | 19 | 9 | 14 | 7
Completed | 18 | 9 | 17 | 7 | 12 | 5
Not Completed | 4 | 2 | 2 | 2 | 2 | 2
Not completed — Adverse Event | 1 | 1 | 1 | 1 | 1 | 0
Not completed — Persistent Positive Blood Cultures | 1 | 0 | 1 | 0 | 0 | 0
Not completed — No relevant bacteria | 2 | 0 | 0 | 0 | 1 | 1
Not completed — Did not receive treatment | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Subject/Parent/Legal Guardian Decision | 0 | 0 | 0 | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Participants who received any dose of IV study medication.
Groups:
- Total: Total of all reporting groups
Arm/Group | Daptomycin - 1 to 6 Year Olds | Comparator- 1 to 6 Year Olds | Daptomycin - 7 to 11 Year Olds | Comparator - 7 to 11 Year Olds | Daptomycin - 12 to 17 Year Olds | Comparator - 12 to 17 Year Olds | Total
Number analyzed (Participants) | 22 | 10 | 19 | 9 | 14 | 7 | 81
Age, Continuous [Mean (Standard Deviation); unit: Years] | 3.81 (1.232) | 4.13 (1.752) | 10.25 (1.217) | 9.46 (1.345) | 14.14 (1.677) | 14.56 (1.868) | 8.70 (4.468)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 8 | 7 | 1 | 0 | 1 | 27
  Male | 12 | 2 | 12 | 8 | 14 | 6 | 54

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With One or More Adverse Events (AEs)
Description: An AE is any untoward medical occurrence in a participant administered a pharmaceutical product that does not necessarily have to have a causal relationship with the treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal product, whether or not related to the medicinal product.
Time Frame: Administration of first dose through the last follow-up visit (up to 77 days)
Population: Participants who received any dose of IV study medication
Measure: Number; unit: Participants
Arm/Group | Daptomycin - 1 to 6 Year Olds | Comparator- 1 to 6 Year Olds | Daptomycin - 7 to 11 Year Olds | Comparator - 7 to 11 Year Olds | Daptomycin - 12 to 17 Year Olds | Comparator - 12 to 17 Year Olds
Number analyzed (Participants) | 22 | 10 | 19 | 9 | 14 | 7
Participants | 15 | 6 | 12 | 9 | 9 | 5

2. Primary Outcome: Number of Participants With One or More Serious Adverse Events (SAEs)
Description: An SAE is any adverse experience occurring at any dose that results in any of the following outcomes: death, life threatening experience, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability or incapacity, is a congenital anomaly or birth defect, or is considered to be an important medical event.
Time Frame: Administration of first dose through the last follow-up visit (up to 77 days)
Population: Participants who received any dose of IV study medication
Measure: Number; unit: Participants
Arm/Group | Daptomycin - 1 to 6 Year Olds | Comparator- 1 to 6 Year Olds | Daptomycin - 7 to 11 Year Olds | Comparator - 7 to 11 Year Olds | Daptomycin - 12 to 17 Year Olds | Comparator - 12 to 17 Year Olds
Number analyzed (Participants) | 22 | 10 | 19 | 9 | 14 | 7
Participants | 6 | 2 | 4 | 3 | 3 | 2

3. Primary Outcome: Percentage of Participants With Maximum Post-Baseline Creatine Phosphokinase (CPK) Elevations Above Upper Limit of Normal
Description: Blood was drawn from baseline up to the end of therapy visit to determine the percentage of participants with maximum post-baseline CPK elevations above the upper limit of 500 Units Per Liter (U/L) .
Time Frame: Baseline up to end of therapy visit (up to 49 days)
Population: Participants who received any dose of IV study medication
Measure: Number; unit: Percentage of Participants
Arm/Group | Daptomycin - 1 to 6 Year Olds | Comparator- 1 to 6 Year Olds | Daptomycin - 7 to 11 Year Olds | Comparator - 7 to 11 Year Olds | Daptomycin - 12 to 17 Year Olds | Comparator - 12 to 17 Year Olds
Number analyzed (Participants) | 22 | 10 | 19 | 9 | 14 | 7
Percentage of Participants | 40.9 | 40.0 | 10.5 | 0.0 | 28.6 | 14.3

4. Primary Outcome: Percentage of Participants With Sustained CPK Elevations
Description: Blood was drawn from baseline up to the end of therapy visit to determine the percentage of participants with sustained CPK elevations, defined as two consecutive post-baseline values above the upper limit of normal (ULN)
Time Frame: Baseline up to end of therapy visit (up to 44 days)
Population: Participants who received any dose of IV study medication
Measure: Number; unit: Percentage of Participants
Arm/Group | Daptomycin - 1 to 6 Year Olds | Comparator- 1 to 6 Year Olds | Daptomycin - 7 to 11 Year Olds | Comparator - 7 to 11 Year Olds | Daptomycin - 12 to 17 Year Olds | Comparator - 12 to 17 Year Olds
Number analyzed (Participants) | 22 | 10 | 19 | 9 | 14 | 7
Percentage of Participants | 18.2 | 20.0 | 0.0 | 0.0 | 28.6 | 14.3

5. Primary Outcome: Number of Participants With Abnormal Focused (Peripheral) Neurological Assessments at Test of Cure (TOC)
Description: Focused neurological examinations were done at the TOC/Safety Visit. These examinations include assessments of sensation, pupillary reflex and tracking, peripheral reflexes (biceps, patellar tendon, ankle jerk and plantar response), muscle tone and strength (upper and lower limbs), coordination (finger to nose) and tremor of the hands/fingers.
Time Frame: TOC Safety Visit (up to 56 days)
Population: Participants who received any dose of IV study medication.
Measure: Number; unit: Participants
Arm/Group | Daptomycin - 1 to 6 Year Olds | Comparator- 1 to 6 Year Olds | Daptomycin - 7 to 11 Year Olds | Comparator - 7 to 11 Year Olds | Daptomycin - 12 to 17 Year Olds | Comparator - 12 to 17 Year Olds
Number analyzed (Participants) | 22 | 10 | 19 | 9 | 14 | 7
Participants
  Alertness | 0 | 0 | 0 | 0 | 0 | 0
  Pupillary Reflex and Tracking | 0 | 0 | 1 | 0 | 0 | 0
  Peripheral Reflex - Biceps | 0 | 0 | 0 | 0 | 0 | 0
  Peripheral Reflex - Patellar Tendon | 0 | 0 | 1 | 0 | 0 | 0
  Peripheral Reflex - Ankle Jerk | 0 | 0 | 1 | 0 | 0 | 0
  Peripheral Reflex - Plantar Response | 0 | 0 | 0 | 0 | 0 | 0
  Muscle Tone - Lower/Upper Limbs | 0 | 0 | 0 | 0 | 2 | 0
  Muscle Strength - Lower/Upper Limbs | 0 | 0 | 0 | 0 | 2 | 0
  Coordination - (Finger to Nose) | 0 | 0 | 0 | 0 | 0 | 0
  Tremor of the hands/fingers | 0 | 0 | 1 | 0 | 0 | 0
  Sensation | 0 | 0 | 0 | 0 | 0 | 0

6. Secondary Outcome: Percentage of Participants With Clinical Success at TOC/Safety Visit
Description: Clinical success was determined by assessing resolution/improvement of signs and symptoms. An assessment of cure or improved is considered clinical success. Cure: resolution of clinically significant signs and symptoms associated with admission infection; no further antibiotic therapy is required for the primary infection under study. Improvement: partial resolution of clinical signs/symptoms of infection such that no further antibiotic therapy is required for the primary infection under study.
Time Frame: 7-14 days after the last dose of study medication (up to 56 days)
Population: All randomized and treated participants who received ≥1 dose of study drug and who had proven S. aureus bacteremia at baseline.
Measure: Number; unit: Percentage of participants
Arm/Group | Daptomycin - 1 to 6 Year Olds | Comparator- 1 to 6 Year Olds | Daptomycin - 7 to 11 Year Olds | Comparator - 7 to 11 Year Olds | Daptomycin - 12 to 17 Year Olds | Comparator - 12 to 17 Year Olds
Number analyzed (Participants) | 20 | 8 | 17 | 9 | 14 | 5
Percentage of participants
  Cured | 80.0 | 87.5 | 94.1 | 77.8 | 78.6 | 60.0
  Improved | 5.0 | 0 | 0 | 0 | 7.1 | 0
Statistical Analysis 1: Comparison: Daptomycin - 1 to 6 Year Olds vs Comparator- 1 to 6 Year Olds; Difference in satisfactory response between treatment groups. Satisfactory response = cured + improved; Test type: Superiority or Other; Difference (%) = -2.5, 95% CI 2-sided [-30.3 to 25.3] — Daptomycin minus Comparator 95% Confidence Interval (CI) by Wilson score method
Statistical Analysis 2: Comparison: Daptomycin - 7 to 11 Year Olds vs Comparator - 7 to 11 Year Olds; Difference in satisfactory response between treatment groups. Satisfactory response = cured + improved; Test type: Superiority or Other; Difference (%) = 16.3, 95% CI 2-sided [-13.0 to 45.7] — Daptomycin minus Comparator 95% CI by Wilson score method
Statistical Analysis 3: Comparison: Daptomycin - 12 to 17 Year Olds vs Comparator - 12 to 17 Year Olds; Difference in satisfactory response between treatment groups. Satisfactory response = cured + improved; Test type: Superiority or Other; Difference (%) = 25.7, 95% CI 2-sided [-21.0 to 72.4] — Daptomycin minus Comparator 95% CI by Wilson score method

7. Secondary Outcome: Percentage of Participants With Overall Success at TOC Visit
Description: Overall success is based on microbiologic responses after initiating study drug and clinical response at TOC/Safety Visit. Overall outcome is a success if both clinical and microbiologic outcomes are successes. An assessment of cure or improved is considered clinical success. Microbiological Success: a participant for whom all baseline infecting pathogens were eradicated (presumed or documented) within 7 days from the start of study drug for uncomplicated bacteremia with no source of infection present, and 10 days for complicated bacteremia or when the source of infection has not been removed.
Time Frame: 7-14 days after the last dose of study medication (up to 56 days)
Population: as for outcome 6
Measure: Number; unit: Percentage of participants
Arm/Group | Daptomycin - 1 to 6 Year Olds | Comparator- 1 to 6 Year Olds | Daptomycin - 7 to 11 Year Olds | Comparator - 7 to 11 Year Olds | Daptomycin - 12 to 17 Year Olds | Comparator - 12 to 17 Year Olds
Number analyzed (Participants) | 20 | 8 | 17 | 9 | 14 | 5
Percentage of participants | 80.0 | 75.0 | 82.4 | 44.4 | 50.0 | 60.0
Statistical Analysis 1: Comparison: Daptomycin - 1 to 6 Year Olds vs Comparator- 1 to 6 Year Olds; Difference in success response between treatment arms; Test type: Superiority or Other; Difference (%) = 5.0, 95% CI 2-sided [-29.8 to 39.8] — Daptomycin minus Comparator 95% CI by Wilson score method
Statistical Analysis 2: Comparison: Daptomycin - 7 to 11 Year Olds vs Comparator - 7 to 11 Year Olds; Difference in success response between treatment arms; Test type: Superiority or Other; Difference (%) = 37.9, 95% CI 2-sided [0.7 to 75.1] — Daptomycin minus Comparator 95% CI by Wilson score method
Statistical Analysis 3: Comparison: Daptomycin - 12 to 17 Year Olds vs Comparator - 12 to 17 Year Olds; Difference in success response between treatment arms; Test type: Superiority or Other; Difference (%) = -10.0, 95% CI [-60.3 to 40.3] — Daptomycin minus Comparator 95% CI by Wilson score method

8. Secondary Outcome: Trough Plasma Concentration of Daptomycin
Description: Plasma concentrations of daptomycin were measured on Days 3 through 6 of IV dosing. Trough concentrations were collected 22 to 26 hours following the end of the previous day's end of infusion and before the next infusion. Concentrations below the limit of quantification were excluded.
Time Frame: Days 3, 4, 5 or 6 of treatment at pre-dose
Population: Participants treated with daptomycin with at least one trough sample. Participants in the comparator treatment groups were not analyzed as they were not treated with daptomycin.
Measure: Mean (Standard Deviation); unit: µg/mL
Arm/Group | Daptomycin - 1 to 6 Year Olds | Comparator- 1 to 6 Year Olds | Daptomycin - 7 to 11 Year Olds | Comparator - 7 to 11 Year Olds | Daptomycin - 12 to 17 Year Olds | Comparator - 12 to 17 Year Olds
Number analyzed (Participants) | 3 | 0 | 10 | 0 | 7 | 0
µg/mL | 4.72 (1.643) |  | 6.39 (3.035) |  | 14.69 (19.109) |

9. Secondary Outcome: Maximum Plasma Concentration (Cmax) of Daptomycin
Description: Plasma concentrations of daptomycin were measured on Days 3 through 6 of IV dosing. Peak concentrations were collected up to 15 minutes following the end of infusion. Concentrations below the limit of quantification were excluded.
Time Frame: Days 3, 4, 5 or 6 of treatment at end of infusion
Population: Participants treated with daptomycin with at least one peak sample. Participants in the comparator treatment groups were not analyzed as they were not treated with daptomycin.
Measure: Mean (Standard Deviation); unit: µg/mL
Arm/Group | Daptomycin - 1 to 6 Year Olds | Comparator- 1 to 6 Year Olds | Daptomycin - 7 to 11 Year Olds | Comparator - 7 to 11 Year Olds | Daptomycin - 12 to 17 Year Olds | Comparator - 12 to 17 Year Olds
Number analyzed (Participants) | 15 | 0 | 18 | 0 | 8 | 0
µg/mL | 96.69 (32.946) |  | 87.66 (34.992) |  | 74.70 (34.909) |

ADVERSE EVENTS:
Time Frame: Administration of first dose through the last follow-up visit (up to 77 days).
Description: Participants who received any dose of IV study medication
Arm/Group | Daptomycin - 1 to 6 Year Olds | Comparator - 1 to 6 Year Olds | Daptomycin - 7 to 11 Year Olds | Comparator - 7 to 11 Year Olds | Daptomycin - 12 to 17 Year Olds | Comparator - 12 to 17 Year Olds
Serious Adverse Events (participants affected / at risk) | 6/22 | 2/10 | 4/19 | 3/9 | 3/14 | 2/7
Other Adverse Events (participants affected / at risk) | 9/22 | 6/10 | 11/19 | 9/9 | 8/14 | 5/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Daptomycin - 1 to 6 Year Olds (N=22) | Comparator - 1 to 6 Year Olds (N=10) | Daptomycin - 7 to 11 Year Olds (N=19) | Comparator - 7 to 11 Year Olds (N=9) | Daptomycin - 12 to 17 Year Olds (N=14) | Comparator - 12 to 17 Year Olds (N=7)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Device breakage (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intestine transplant rejection (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arthritis bacterial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bacteraemia (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bone abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Muscle abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Osteomyelitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Staphylococcal bacteraemia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic enzyme increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malnutrition (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bone fistula (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Synovitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Venous thrombosis limb (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Daptomycin - 1 to 6 Year Olds (N=22) | Comparator - 1 to 6 Year Olds (N=10) | Daptomycin - 7 to 11 Year Olds (N=19) | Comparator - 7 to 11 Year Olds (N=9) | Daptomycin - 12 to 17 Year Olds (N=14) | Comparator - 12 to 17 Year Olds (N=7)
Abdominal lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Thrombocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Ventricular extrasystoles (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 4 (4) | 1 (1) | 1 (1) | 3 (3) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 2 (4) | 2 (4) | 0 (0) | 2 (2) | 0 (0)
Catheter site discharge (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Catheter site oedema (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Catheter site pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Device breakage (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infusion site pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 2 (3) | 1 (1) | 1 (1) | 2 (3) | 2 (2) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Abdominal abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthritis bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Candida infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Infected skin ulcer (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lung abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Osteomyelitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Osteomyelitis acute (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Postoperative wound infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash pustular (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rhinovirus infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Systemic candida (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Varicella (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Excoriation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Wound (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wound dehiscence (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood creatine phosphokinase increased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Blood potassium decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood sodium decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hepatic enzyme increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Transaminases increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Fluid overload (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hypernatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperphosphataemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Myositis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lethargy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abnormal behaviour (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Renal failure acute (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Renal necrosis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Epididymal cyst (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pharyngeal ulceration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash macular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Phlebitis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Thrombophlebitis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Body temperature increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No